CLINICAL TRIAL: NCT02695030
Title: MicroVention Low-profile Visualized Intraluminal Support (LVIS*) or LVIS Jr Humanitarian Use Device (LVIS HUD)
Brief Title: Low-profile Visualized Intraluminal Support -HUD
Status: Approved for marketing | Type: Expanded Access
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 14-01582; 09-0222 (Other: Humanitarian Use Device Designation Number); H130005 (Other: Humanitarian Device Exemption Number)
Record Dates: First submitted 2016-02-24; First posted 2016-03-01 (Estimated); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Giant Wide Necked Aneurysms

INTERVENTIONS:
Device: Low Profile Visualized Intraluminal Support Device — LVIS device is intended for use with bare platinum embolic coils for the treatment of unruptured, wide neck, intracranial, saccular aneurysms.
  Other Names: Intracranial Stent

SUMMARY:
The MicroVention Low-profile Visualized Intraluminal Support (LVIS*) Device is intended for use with bare platinum embolic coils for the treatment of unruptured, wide neck (neck greater than or equal to 4 or a dome to neck ratio less than two), intracranial, saccular aneurysms arising from a parent vessel with a diameter of greater than or equal to 2.5mm and less than or equal to 4.5mm.

DETAILED DESCRIPTION:
Wide neck aneurysms are very difficult to treat both surgically and endovascularly with clipping or coiling. The availability of this neurovascular flow diverter as a Humanitarian Use Device has provided an additional approach to aneurysm occlusion using endovascular techniques.

ELIGIBILITY:
Inclusion Criteria:

* Wide neck (neck greater than or equal to 4 or a dome to neck ratio less than two),Intracranial, saccular aneurysm arising from a parent vessel with a diameter of greater than or equal to 2.5mm and less than or equal to 4.5mm.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Howard Riina, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States